CLINICAL TRIAL: NCT04124627
Title: Place of Ultrasound Guidance of Surgery Site in Surgery for Lumbar Canal Stenosis and Lumbar Disc Herniations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Medico-Chirurgicale et Obstetrique Cote d'Opale (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ULTRALUMBAR
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Lumbar Stenosis, Familial
Keywords: Ultrasound guidance; surgery for lumbar spine; irradiation; wrong site surgery
MeSH Terms: conditions — Lumbar Stenosis, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): Ultrasound plus radiographic guidance
  Interventions: Procedure: Ultrasound guidance in addition to radiographic guidance

INTERVENTIONS:
Procedure: Ultrasound guidance in addition to radiographic guidance — Patients that will be operated will receive ultrasound guidance in addition to radiographic guidance, that is gold standard

SUMMARY:
The identification of the operative site of lumbar ductal stenosis and lumbar disc herniation is classically done by radioscopy, thus inducing irradiation of the patient.

The use of ultrasound in spine surgery is little studied and poorly mentioned in the scientific literature. However, it is commonly used for other types of scouting (especially anesthetics). Thus, in the absence of consensus and clear recommendations, some practitioners perform ultrasound scans . Methodological developments also validate the feasibility of the ultrasound approach.

The double benefit of an ultrasound identification is firstly a lack of exposure to X-rays for both the patient and the operating team and secondly a lower cost than a conventional radiography.

The main objective is to demonstrate the interest of the ultrasound identification of the surgical site in the intervention of lumbar ductal stenosis and lumbar disc herniations in terms of concordance of the operating site between ultrasound and fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Patients who gave their consent
* Patients requiring surgery for the treatment of lumbar stenosis or lumbar disc herniation

Exclusion Criteria:

* Pregnant or lactating women according to article L1121-5 of the CSP.
* Vulnerable persons according to article L1121-6 of the CSP.
* Major persons placed under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
concordance of the operating site after radiological and ultrasound guidance | day 1
  ok / not ok

SECONDARY OUTCOMES:
number of shots made and preventable | day 0
  number
preventable radiation dose | day 0
  Gys
exam costs (based on national cost scale) | day 0
  euros

CONTACTS AND LOCATIONS:
Locations (1):
- Centre MCO Côte d'Opale, Boulogne-sur-Mer, Pas De Calais, France